CLINICAL TRIAL: NCT04040452
Title: Continuous Infusion Versus Intermittent Ketorolac for Postoperative Pain Control in Pediatric Cardiac Surgery Patients
Brief Title: Continuous vs Intermittent Ketorolac for Pain Control in Peds CV Surgery
Acronym: CIVIK
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Phoenix Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 166166
Record Dates: First submitted 2019-07-29; First posted 2019-07-31 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-02

CONDITIONS: Congenital Heart Disease in Children
Keywords: pain control; cardiac surgery; pediatric; opioid; NSAID; congenital heart disease
MeSH Terms: conditions — Agnosia; Heart Defects, Congenital

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): 1. Description: Patients randomized for the treatment arm of the study group will receive a continuous infusion of ketorolac plus an intermittent dose of placebo (plasmalyte). To eliminate excess exposure and the associated side effects, all patients enrolled in the study will not be given any additional NSAIDs (except aspirin, which is standard of care in many post-operative cardiac surgery patients) during the study period.
  2. Dosage and Route of Administration:
     1. Continuous ketorolac 0.08mg/kg/hr, with a maximum of 5mg/hr for patients weighing greater than or equal to 60kg, administered intravenously by nursing staff. Study drug will infuse continuously for 48 hours.
     2. Intermittent Plasmalyte 0.033mL/kg (max 2mL) infusion every 6 hours for 48 hours.
  Interventions: Drug: Continuous ketorolac
- Standard of care (Placebo Comparator): 1. Description: Patients randomized to the standard of care arm of the study will receive a generically marked syringe of Plasmalyte to be infused at the same rate as the treatment medication, and will only receive intermittent dosing of ketorolac (current standard of care). As in the treatment group, no additional NSAIDs (except aspirin) are to be given during the 48 hour study period.
  2. Dosage and Route of Administration
     1. Continuous Plasmalyte infusion to match the aforementioned ketorolac dosing
     2. Intermittent ketorolac 0.5mg/kg IV infusion every 6 hours (max 30mg per dose)
  Interventions: Drug: Continuous ketorolac

INTERVENTIONS:
Drug: Continuous ketorolac — Patients randomized for the treatment arm of the study group will receive a continuous infusion of ketorolac plus an intermittent dose of placebo (plasmalyte) for 48 hours.

SUMMARY:
The proposed study will be a prospective, randomized, double blind, placebo controlled trial to compare the use of a continuous infusion versus intermittent ketorolac on postoperative patients in the pediatric cardiovascular ICU. We intend to determine if the continuous infusion leads to a decreased utilization of opiates when compared to intermittent ketorolac.

DETAILED DESCRIPTION:
The mainstay of postoperative pain control in the CVICU remains opiate-based therapy. Reliance on this class of medications can be detrimental, contributing to complications including hemodynamic instability, dependency, and withdrawal which can ultimately lead to longer hospital admissions, as well as long term and persistent neurodevelopmental effects. In addition, the opioid crisis has driven practitioners to aim for methods to reduce opioid exposure and post-operative narcotic prescriptions in pediatric and adult patients alike. There is a growing body of evidence in the adult literature showing promising results with the use of a continuous infusion of ketorolac in postoperative patients, including in a pediatric population. What the current literature has failed to show is whether a continuous infusion of ketorolac post operatively decreases the use of opiate mediations in a pediatric population compared to intermittent bolus injections, which is the current standard of care. Given the sensitivity and fragility inherent in those patients with CHD, working to reduce deleterious effects from excessive and prolonged opiate exposure is imperative. This study aims to examine whether the use of a continuous infusion of ketorolac can reduce the amount of opiates needed to treat postoperative pain control in the pediatric CVICU population, in comparison to patients who receive intermittent ketorolac within the first 72 hours post-operatively.

ELIGIBILITY:
Inclusion Criteria:

1. All patients aged 3 months to 4 years 11months admitted post operatively to the CVICU during the time period in which the study will be ongoing
2. Initiation of study medication within the first 12-24 hours post-operatively
3. The cardiovascular attending of record after review of the intraoperative course and post-operative laboratories determines the patient will receive Ketorolac for pain control

Exclusion Criteria:

1. Patients that have acute kidney injury, as defined by the letter "I" in the pRIFLE criteria.
2. History of allergy or sensitivity reaction to ketorolac or any NSAID medications.
3. Requiring mechanical circulatory support (ECMO) or continuous renal replacement therapy (CRRT) within the first 48 hours post-operatively
4. Orthotopic heart transplantation
5. Clinically significant bleeding
6. Patients with known pre-operative medical renal disease, renal transplantation history, congenital or acquired renal abnormality or deformity

Ages: 3 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 166 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
1. Total fentanyl dose equivalents received within the first 96 hours post-operatively | Within 72 hours of cardiac surgery
  The total opioid receipt (converted to fentanyl equivalents) administered to patients enrolled in the study within the first 96 hours after cardiac surgery.

SECONDARY OUTCOMES:
1. Total fentanyl equivalents received in each 24 hour period before and after initiating the study drug | Within 72 hours after cardiac surgery
  The total opioid receipt (converted to fentanyl equivalents) administered to patients enrolled in the study within each 24 hour period after cardiac surgery (up to 96 hours post-operatively).
Rate of acute kidney injury measured by pRIFLE criteria | Within 72 hours after cardiac surgery
  Acute kidney injury rates
Major bleeding events | Within 72 hours after cardiac surgery
  Hemoglobin decrease > 2 g/dL, requirement of 2 or more units of PRBC's/whole blood, or development of symptomatic/clinically evident bleeding in any organ or compartment
Pain scores | Within 72 hours after cardiac surgery
  FLACC scores (face, legs, activity, cry, consolability): score of 0-10 (10 being most severe pain, 0 being least severe). 0 = relaxed/comfortable, 1-3 = mild discomfort, 4-6 = moderate pain, 7-10 = severe discomfort or pain or both
Sedative agent requirements | Within 72 hours after cardiac surgery
  Dose receipt/drug selection of sedative agents

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Engelhardt, MD, Principal Investigator — Heart Center
Locations (1):
- Phoenix Children's Hospital, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to make IPD available to other researchers.

REFERENCES:
- [Background] Onaka T, Yagi K. Differential effects of naloxone on neuroendocrine responses to fear-related emotional stress. Exp Brain Res. 1990;81(1):53-8. doi: 10.1007/BF00230100. PMID 2168320
- [Background] Burd RS, Tobias JD. Ketorolac for pain management after abdominal surgical procedures in infants. South Med J. 2002 Mar;95(3):331-3. PMID 11902701
- [Background] Burns JW, Aitken HA, Bullingham RE, McArdle CS, Kenny GN. Double-blind comparison of the morphine sparing effect of continuous and intermittent i.m. administration of ketorolac. Br J Anaesth. 1991 Sep;67(3):235-8. doi: 10.1093/bja/67.3.235. PMID 1911008
- [Background] Cohen MN, Christians U, Henthorn T, Vu Tran Z, Moll V, Zuk J, Galinkin J. Pharmacokinetics of single-dose intravenous ketorolac in infants aged 2-11 months. Anesth Analg. 2011 Mar;112(3):655-60. doi: 10.1213/ANE.0b013e3182075d04. Epub 2011 Jan 13. PMID 21233498
- [Background] Dawkins TN, Barclay CA, Gardiner RL, Krawczeski CD. Safety of intravenous use of ketorolac in infants following cardiothoracic surgery. Cardiol Young. 2009 Feb;19(1):105-8. doi: 10.1017/S1047951109003527. Epub 2009 Jan 12. PMID 19134246
- [Background] Grimsby GM, Conley SP, Trentman TL, Castle EP, Andrews PE, Mihalik LA, Hentz JG, Humphreys MR. A double-blind randomized controlled trial of continuous intravenous Ketorolac vs placebo for adjuvant pain control after renal surgery. Mayo Clin Proc. 2012 Nov;87(11):1089-97. doi: 10.1016/j.mayocp.2012.07.018. Epub 2012 Oct 8. PMID 23058854
- [Background] Gupta A, Daggett C, Drant S, Rivero N, Lewis A. Prospective randomized trial of ketorolac after congenital heart surgery. J Cardiothorac Vasc Anesth. 2004 Aug;18(4):454-7. doi: 10.1053/j.jvca.2004.05.024. PMID 15365927
- [Background] Howard ML, Isaacs AN, Nisly SA. Continuous Infusion Nonsteroidal Anti-Inflammatory Drugs for Perioperative Pain Management. J Pharm Pract. 2018 Feb;31(1):66-81. doi: 10.1177/0897190016665539. Epub 2016 Aug 31. PMID 27580638
- [Background] Britton J, Martinez FD. The relationship of childhood respiratory infection to growth and decline in lung function. Am J Respir Crit Care Med. 1996 Dec;154(6 Pt 2):S240-5. doi: 10.1164/ajrccm/154.6_Pt_2.S240. No abstract available. PMID 8970395
- [Background] Inoue M, Caldarone CA, Frndova H, Cox PN, Ito S, Taddio A, Guerguerian AM. Safety and efficacy of ketorolac in children after cardiac surgery. Intensive Care Med. 2009 Sep;35(9):1584-92. doi: 10.1007/s00134-009-1541-1. Epub 2009 Jun 27. PMID 19562323
- [Background] Jalkut MK. Ketorolac as an analgesic agent for infants and children after cardiac surgery: safety profile and appropriate patient selection. AACN Adv Crit Care. 2014 Jan-Mar;25(1):23-30; quiz 31-2. doi: 10.1097/NCI.0000000000000002. PMID 24441450
- [Background] Moffett BS, Wann TI, Carberry KE, Mott AR. Safety of ketorolac in neonates and infants after cardiac surgery. Paediatr Anaesth. 2006 Apr;16(4):424-8. doi: 10.1111/j.1460-9592.2005.01806.x. PMID 16618297